CLINICAL TRIAL: NCT02953158
Title: A Comparison of A Hypocaloric Diet Plus One Hass Avocado Per Day Versus An Equally Hypocaloric Diet for Weight Loss, Satiety, Changes in Body Composition, and Risk Factors for Chronic Disease (HAWLS)
Brief Title: Effectiveness of Changing Dietary Fat on Weight Loss
Acronym: HAWLS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Hass Avocado Board (Other)
Responsible Party: Principal Investigator, Zhaoping Li, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB#16-001157
Record Dates: First submitted 2016-10-06; First posted 2016-11-02 (Estimated); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Overweight
MeSH Terms: conditions — Overweight | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Haas Avocado (Experimental): Haas Avocado commercially available Behavioral: Dietary recommendations Recommendation: a hypocaloric weight loss diet
  Interventions: Other: Haas Avocado
- Dietary Counseling (Active Comparator): Behavioral: Dietary Counseling Recommendation: equally hypocaloric usual American diet.
  Interventions: Behavioral: Dietary Counseling

INTERVENTIONS:
Other: Haas Avocado — Hypocaloric weight loss diet
  Other Names: Avocado
  Arms: Haas Avocado
Behavioral: Dietary Counseling — Dietary Counseling
  Arms: Dietary Counseling

SUMMARY:
This study will compare two energy reduced diets; one diet will include one Haas avocado/day while the other diet will follow the usual American dietary pattern. All subjects will receive a dietary plan that reduces their usual intake by 500kcal/day with the same percentage of fat, protein and carbohydrates. The results from this study may help to explain if eating one Haas avocado/day can achieve at least equivalent weight loss when compared to the usual American diet.

DETAILED DESCRIPTION:
Overweight and obesity in the United States and other industrialized countries represents a significant and growing health problem. Individuals who are overweight or obese increase their risk of coronary heart disease (CHD), diabetes (T2D), and the metabolic syndrome. Obesity affects both genders and every ethnicity in the United States. The prevalence of obesity in the United States is currently 32.2% in adult men and 35.5% in adult women. The most recent evidence indicates that 33.8% of adults, over 66 million American adults, are obese (30 million men and 36 million women) while an additional 74 million (42 million men and 32 million women) are overweight. The prevalence of obesity has grown a shocking 40% over the last 30 years.

These problems are truly global in nature. In European countries obesity ranges from 20-30% of the population and is even higher in Australia, South America, and Polynesia. The World Health Organization estimates that there will be over 1.5 billion obese individuals worldwide by 2020 if current trends continue.

Calorie controlled diets have routinely been demonstrated to help in both short and long-term weight reduction in individuals who are overweight or obese. In particular, hypocaloric diets, with a calorie reduction of 500 kcals per day have been shown in numerous studies to result in safe and effective weight loss.

It is important for individuals who are following weight loss programs to maintain healthy nutritional patterns, to maintain or improve their dietary quality. Haas avocados can play a significant role as part of a healthy weight loss program and help individuals not only improve their dietary quality, but also lower their risk of chronic diseases such as CHD, T2D, and the metabolic syndrome. Avocados are high in monounsaturated fat, dietary fiber, and a variety of other important phytochemicals such as lutein, vitamin E, niacin and folate. Despite these multiple nutritional benefits, myths exist that avocados may be fattening due to their fat and calorie content and therefore, should be avoided by people trying to lose weight.

The current research trial is designed to compare two energy reduced (hypocaloric) diets. One diet will include one Hass avocado/day, while achieving a 500 kcal/day energy reduction. The other diet will follow a usual American diet pattern, but will also include an energy restriction of 500 kcals/day. Parameters to be explored include weight loss, satiety, dietary quality, changes in body composition and risk factors for chronic disease.

ELIGIBILITY:
Inclusion Criteria:

Male or female between the ages of 20-60 years of age.

* Body Mass Index (BMI) 27.0 -35.0 kg/m2.
* Not currently taking a prescription medication for weight loss (e.g. orlistat (Xenical®), sibutramine (Meridia®) or phentermine etc.) If subject is willing to discontinue prescription medication(s) immediately and willing to refrain from taking medication(s) for duration of study, he/she may be enrolled after a four-week washout period.
* Not currently taking any over-the-counter weight loss supplement(s) or appetite suppressants (including OTC stimulants). If subject is willing to discontinue supplement(s) immediately and willing to refrain from taking supplement(s) for duration of study, he/she may be enrolled after a two-week washout period.
* Not currently enrolled in any commercial weight loss program (e.g. Jenny Craig, Weight Watchers), internet based weight-management program, self-help group (e.g. TOPS, Overeaters Anonymous) or participating in any food preparation/delivery program (eg Nutrisystems). If subject is willing to discontinue program immediately and willing to refrain from program for duration of study, he/she may be included after a two-week washout period.
* Willing to keep and turn in a daily log/compliance book as required by study protocol.
* Willingness and ability to make all scheduled appointments.
* Willing to follow dietary recommendations required by study protocol.
* Willingness to complete Dual X-Ray Absorptiometry (DXA) procedure.
* Willingness to periodically have small blood samples drawn as indicated in the protocol.

Exclusion Criteria:

More than a 5 pound weight gain or weight loss within the 3 months prior to enrollment in the study.

* History of thyroid disease, but not taking medication or medication dosage changed one or more times over last 6 months. History of thyroid disease and on a stable dose of prescription medication for 6 months or longer is acceptable.
* Diagnosed with Type I or Type II diabetes. History of major surgery within three months of enrollment.
* History of heart problems (e.g. angina, bypass surgery, MI, etc.) within three months prior to enrollment.
* Presence of implanted cardiac defibrillator or pacemaker.
* Uncontrolled hypertension/high blood pressure.
* History of a surgical procedure for weight loss at any time (e.g. gastroplasty, gastric by-pass, gastrectomy or partial gastrectomy).
* Gastrointestinal disorders including chronic malabsorptive conditions, peptic ulcer disease, Crohn's disease, chronic diarrhea or active gallbladder disease.
* History of inflammatory bowel disease.
* Following a diet that requires the elimination of FODMAPS•
* Following a specific diet that restricts specific food groups (eg. Paleo) or with extreme macronutrient ratios (carbohydrates, fats and proteins). • History of fatty liver.
* History or presence of cancer. Persons with successfully resected basal cell carcinoma of the skin may be enrolled if treatment completed more than 6 months prior to enrollment.
* History of clinically diagnosed eating disorders including anorexia nervosa, bulimia nervosa or binge eating disorder.
* Women who are pregnant, lactating or trying to become pregnant.
* Currently taking any prescription medication for less than 3 months.
* Currently taking any prescriptions drugs that may impact weight regulation
* Currently consuming >14 alcoholic drinks (1 drink = 12 fl oz beer, 4 fl oz wine or 1.5 fl oz liquor) per week and/or unwilling to limit intake to less than 3 drinks per week during study participation.
* Known allergy to avocados.
* History of alcohol dependency.
* Participation in another clinical trial within 30 days prior to enrollment.
* Currently smoking cigarettes.
* Any clinically significant food allergy.
* Currently consuming an average of >1 avocado per week.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Change in weight loss after consumption of 1 Haas Avocado per day with a hypocaloric diet | Baseline to 12 weeks
  Individuals will be randomly assigned to a hypocaloric (500 Cal deficit) meal plans with or without one Hass avocado a day for 12 weeks.

SECONDARY OUTCOMES:
Change in gut microbiome | Baseline to 12 weeks
  Individuals will be randomly assigned to a hypocaloric (500 Cal deficit) meal plans with or without one Hass avocado a day for 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoping Li, MD, PhD, Principal Investigator — UCLA Center for Human Nutrition
Locations (1):
- UCLA Center for Human Nutrition, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Henning SM, Yang J, Woo SL, Lee RP, Huang J, Rasmusen A, Carpenter CL, Thames G, Gilbuena I, Tseng CH, Heber D, Li Z. Hass Avocado Inclusion in a Weight-Loss Diet Supported Weight Loss and Altered Gut Microbiota: A 12-Week Randomized, Parallel-Controlled Trial. Curr Dev Nutr. 2019 Jun 12;3(8):nzz068. doi: 10.1093/cdn/nzz068. eCollection 2019 Aug. PMID 31367691